CLINICAL TRIAL: NCT06508853
Title: Exploring the Experience of Support Workers and Managers Supporting People With Learning Disabilities Who Have Moved From Inpatient to Community Settings as Part of the Transforming Care Agenda.
Brief Title: Transforming Care Experiences of Support Workers and Managers
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 339318
Record Dates: First submitted 2024-07-15; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Learning Disabilities; Behavioural Problem
MeSH Terms: conditions — Learning Disabilities; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative research (no intervention) — Interviews are being conducted with support workers and managers.

SUMMARY:
* What research question is being addressed? What is the experience of support workers, and managers, supporting people with learning disabilities who have moved from inpatient to community settings as part of the Transforming Care Agenda.
* How is it of relevance and importance to patients and public? In 2011 serious abuse of people with learning disabilities was uncovered at Winterbourne View, an independent hospital for people with learning disabilities. The Transforming Care Agenda was set out by the UK government in 2012 in response to this abuse. A key part of the action plan included moving people with learning disabilities out of inappropriate hospital settings, into the community.

Support workers and managers are key mediators in approaches to ensure that people with learning disabilities are able to achieve a good quality of life in the community, however so far there is limited research looking into their experiences.

* Broadly what area (disease, therapy or service) is being studied? For therapeutic studies what is the drug, device or procedure being tested? The area being studied is support for people with learning disabilities who have moved from inpatient settings to community settings.
* Who would be eligible? Support workers and managers who have worked with people with learning disabilities who have moved from inpatient to community settings within the past three years will be eligible to be interviewed as part of this study. 4 to 6 support workers, and 4 to 6 managers will be interviewed in total.
* The type of sites where the study will be conducted Participants (support workers and managers) will be recruited through NHS sites (community learning disability teams) who have identified individuals with learning disabilities who have moved from hospital to community settings (as part of the Transforming Care Agenda) within the past 3 years.
* How long will the study last and what will the participants undergo? The study will last approximately 1.5 years. If they consent, participants will be invited to take part in an interview, lasting up to one hour. The interview will focus on their experience of supporting someone with a learning disability who has moved from a hospital setting, into a community setting, within the past three years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be support workers and managers working within services for people with learning disabilities (supported living or care home settings).
2. Participants need to have worked with someone who has a learning disability who has been discharged from hospital during the past three years.
3. Participants need to have worked with the person with a learning disability during the first three years of their discharge from hospital.
4. Participants need to have worked with the person who has a learning disability for a period of at least four months.
5. The person with a learning disability will need to have been discharged from hospital, into their current service, within the past 3 years.
6. For each person with a learning disability identified, a maximum of two support workers and one manager can be included (interviewed).
7. Support workers or managers will need to be based within one of the four research site localities (South London and Maudsley, Hertfordshire NHS University Trust, East London Foundation Trust and North East London Foundation Trust).
8. Support workers and managers will need to be able to participate in interviews on Microsoft Teams, or in person, conducted in the English language.
9. There are no inclusion or exclusion criteria based on age, gender, ability or any other personal identifiers.

Exclusion Criteria:

1. Support workers or managers working with autistic people, or people who have experienced mental health difficulties (without a learning disability).
2. Support workers or managers who have worked with the person with a learning disability for less than four months.
3. Support workers or managers working in locations outside of the remit of any of the four research sites.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be support workers and managers working with people with learning disabilities who have moved from hospital to community settings as part of the transforming care agenda.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
No formal outcome measures - qualitative analysis of data from interviews. | 1
  Data will be analysed using IPA

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No